CLINICAL TRIAL: NCT02834091
Title: Satisfaction Survey of Patients Over Hypnoanalgesia or Hypnosedation at a Digestive Endoscopy or Surgery
Acronym: SEDuCE
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: SEDuCE
Record Dates: First submitted 2016-06-30; First posted 2016-07-15 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Endoscopy; Surgery, Digestive System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Hypnoanalgesia

SUMMARY:
The use of hypnosedation in the context of anesthesia is validated. This is a technique that combines the hypnosis procedure as intravenous sedation. For surgery, it is associated with local anesthesia surgical site. It can favorably replace general anesthesia if surgery or endoscopy allows but doctors will always need local anesthesia surgical site where surgery The hospital Paris Saint joseph introduced gradually this technique from first in 2007 to the operating room and in the various services of conventional and ambulatory hospitalizations.

The goal of the investigators is to evaluate these parameters on a prospective cohort of patients supported by hypnosedation in Paris Saint Joseph hospital for an endoscopy or surgery.

DETAILED DESCRIPTION:
The use of medical hypnosis has been developing for about fifteen years in several health facilities.

The Hospital Group Paris Saint-Joseph has progressively introduced first this technique from 2007 to the operating room and in the various services of conventional and ambulatory hospitalizations.

The French Society of Anesthesia and Intensive Care (SFAR) recognizes the hypnosedation as sedation technique that can be used in acute pain and anesthesia (operating theater, emergency, painful treatments ...).

There are currently many quality scientific papers published in international journals in particular by the team of Pr. M. E. Faymonville Liege, who explained the mechanisms and consequences of hypnosedation.

The use of hypnosedation in the context of anesthesia is validated. This is a technique that combines the hypnosis procedure as intravenous sedation. For surgery, it is associated with local anesthesia surgical site. It can favorably replace general anesthesia if surgery or endoscopy allows but doctors will always need local anesthesia surgical site where surgery. It can also complement a regional anesthesia to increase patient comfort (less stress, anxiety and pain) .If necessary, the conversion of general anesthesia hypnosedation is always possible during surgery or gastrointestinal endoscopy.

In the Paris Saint joseph Hospital facility, several anesthesiologists and nurse anesthetists are trained in medical hypnosis. Now, a common practice in surgery hypnosedation (inguinal hernia, thyroid and para-thyroid surgery) and endoscopy (colonoscopy, gastroesophageal gastroduodenal endoscopy) .On a period of 3 years, 414 acts were carried out under hypnosedation. When digestive endoscopy adding sedation is not systematic and, if the patient is comfortable enough without conscious sedation, only hypnoanalgesia is used (use of hypnosis in the prevention or relief of acute pain or chronic).

This technique is part of the panel modes of analgesia and anesthesia can be offered to patients. However, little is known about patient satisfaction and their experiences during the procedure under hypnosedation.

The objective is to evaluate these parameters on a prospective cohort of patients supported by hypnosedation in Paris Saint Joseph hospital for an endoscopy or surgery.

This evaluation is part of the evaluation of professional practices (EPP) recommended by the HAS (french High Authority of Health) and the ARS (Regional Health Agency).

Main objective / secondary

Primary objective :

Measure satisfaction of patients resorted to hypnosedation or hypnoanalgesia during an endoscopy or surgery

Secondary objective:

Measure the doses of drugs used for conscious sedation

Methodology :

* DESIGN: Prospective cohort single-center, non-interventional kind EPP on the satisfaction of patients who underwent hypnosedation for surgery or endoscopy
* Duration of the study: 8 months (November 2015-June 2016): the estimated number of 80 patients
* Acquisition of data:
* Age, weight, height, gender, ASA (Physical status score) score
* Type of surgery or endoscopy
* Previous history of surgery or endoscopy
* Names and doses of treatments
* Conversion to general anesthesia yes / no
* Length of management in operating room
* Adverse events during surgery and in recovery
* Evaluation using a numerical scale from 0 to 10:
* Patient anxiety during the pre- and per-interventional
* The per-Interventional Pain, Interventional immediate post-and before the release of the SSPI (The post-interventional surveillance room)
* The feeling of active participation in the intervention
* The quality of the relationship with the hypnotist during surgery
* Overall satisfaction during surgery
* Acceptance or not the patient to repeat surgery or examination under the same terms
* Acceptance or not to recommend the patient to the relatives hypnosedation
* Case open for any comments or suggestions obviousness

ELIGIBILITY:
Inclusion Criteria:

* Patients who chose surgery or endoscopy under hypnosedation
* Selected in consultation surgery or gastroenterology for a realization of the act under hypnosedation.
* Having a pre-hypnosedation anesthesia consultation by an anesthesiologist trained in hypnosis with validation of eligibility for hypnosedation.
* No opposition to participate in the study

Exclusion Criteria:

* Absence affiliate to a social security scheme
* Patients not eligible for hypnosedation:
* No specific consultation pre-anesthesia hypnosedation
* Poor understanding of the French language
* Major Hearing problems
* Severe cognitive or psychiatric disorders
* Insufficient reasoning or refusal with respect to the use of hypnosedation
* Administration of anxiolytic premedication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who used the hypnosedation or hypnoanalgesia during an endoscopy or surgery
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2016-01-22 (Actual); Primary Completion 2016-11-02 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Assessment of Patient satisfaction | Day 1 After Hypnoanalgesia or Hypnosedation
  Patient satisfaction rated on a scale from 0 (dissatisfied) to 10 (extremely satisfied).
  An average value:
  * <5: low satisfaction
  * From 5 to 7.4: Average satisfaction •> 7.5: Important satisfaction

SECONDARY OUTCOMES:
Pain Assessment | Day 1 within the first hour after Hypnoanalgesia or Hypnosedation
  Pain:
  An average value:
  * <3: low or no pain
  * From 3 to 5.9: moderate pain •> 5.9: strong pain
Anxiety assessment | Day 1 within the first hour after Hypnoanalgesia or Hypnosedation
  An average value:
  * <3: low or absent anxiety
  * From 3 to 5.9: moderate anxiety •> 5.9: high anxiety

CONTACTS AND LOCATIONS:
Overall Officials: GORY Christian, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No